CLINICAL TRIAL: NCT07082088
Title: Effect of Abutment Hydrophilicity on Soft Tissue Morphogenesis: Histological CCT
Brief Title: Abutment Hydrophilicity on Soft Tissue Morphogenesis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Paolo Pesce (Other)
Responsible Party: Sponsor-Investigator, Paolo Pesce, Professor, Universita degli Studi di Genova
Organization: Universita degli Studi di Genova (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: hydrophilicity
Record Dates: First submitted 2025-06-22; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Missing Tooth/Teeth
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treated abutments (Experimental): abutment allocated to the test group were placed in an Argon plasma reactor (Plasmapp, South Korea) for decontamination and activation
  Interventions: Device: the test group were placed in an Argon plasma reactor
- Non treated abutment (No Intervention): Abutment without any surface treatment

INTERVENTIONS:
Device: the test group were placed in an Argon plasma reactor — the test group were placed in an Argon plasma reactor
  Arms: Treated abutments

SUMMARY:
The goal of this clinical trial is to evaluate the effect of abutment surface bioactivation via argon plasma treatment on peri-implant soft tissue healing and integration in adult patients undergoing implant therapy.

The main questions it aims to answer are:

Does argon plasma treatment of healing abutments improve the quality and organization of peri-implant connective tissue compared to untreated abutments?

Does the treatment influence histological parameters such as epithelial regeneration, vascularization, inflammatory infiltrate, and keratin layer thickness?

Researchers will compare plasma-treated healing abutments to untreated machined-surface abutments to determine whether the bioactivated surface improves soft tissue morphogenesis.

Participants will:

Undergo implant placement with immediate connection of either a treated or untreated healing abutment.

Have plaque and bleeding indices recorded at 3 months.

Undergo a soft tissue biopsy at 3 months for histological analysis (including evaluation of inflammation, connective tissue, epithelial morphology, vascularization, and keratinization).

ELIGIBILITY:
Inclusion Criteria:

* presence of at least 4 mm of keratinized mucosa around the implants
* patients aged 18 years or older
* medically healthy patients (ASA I), or patients with mild systemic disease (ASA II)
* partially edentulous state
* healthy periodontal condition (also including periodontal health on reduced periodontium) according to the referent case definition

Exclusion Criteria:

* ASA physical status 3
* severe smokers (> 10 cig/day)
* patients undergoing bisphosphonate therapy
* pregnant or lactating women
* estrogen-related hormonal disorders or hormonal substitution therapy
* untreated periodontitis (pocket depth 4mm with positive bleeding on probing)
* multiple gingival recession
* patients with a history of head and neck cancers and radiotherapy in this region.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Perimplant tissue inflammation | 3 months after implant insertion
  Evaluation of density and distribution of inflammatory cells (lymphocytes, plasma cells, granulocytes, macrophages) in the peri-epithelial connective tissue will be evaluated and a score will be used; 0 Massive infiltrate, diffusely present throughout the section; dense cellular aggregates; severely disturbed connective architecture.
  1. Intense infiltrate, present in most of the section but not fully diffuse; clearly visible focal aggregates.
  2 Moderate infiltrate, 3 Minimal infiltrate; isolated low-density cellular foci; connective tissue mostly unaffected.
  4 No recognizable inflammatory infiltrate; only resident normal cells present.

SECONDARY OUTCOMES:
Connective tissue maturation | 3 months after implant insertion
  Organization and maturation of collagen fibers in the subepithelial connective tissue. Score:
  0 Immature, disorganized tissue; sparse, wavy, randomly oriented collagen fibers; abundant amorphous matrix; numerous active fibroblasts.
  1. Partial organization: more collagen fibers but still irregularly arranged; thin, wavy fibers; abundant amorphous matrix persists.
  2. Intermediate organization: initial fiber parallelism; collagen bundles alternating with matrix; fibers still partially wavy.
  3. Well organized: parallel collagen bundles along the epithelial plane; reduced interstitial spaces; reduced amorphous matrix; fewer fibroblasts.
  4. Complete maturation: dense, regular collagen bundles; consistent and continuous orientation; dense, stable, poorly cellular connective tissue.
Epithelial regeneration | 3 months after implant insertion
  Evaluation of thickness, continuity, and maturation of the overlying epithelium.
  Scores:
  0 Epithelium absent or severely discontinuous; ulcerated or completely denuded areas.
  1. Partial regeneration: covered zones alternating with denuded or de-epithelialized areas.
  2. Almost complete: continuous epithelium but with reduced thickness and/or not fully stratified cellular structure.
  3. Complete but thin: stratified epithelium present, with fewer cell layers than normal.
  4. Complete, stratified epithelium; well-developed with multiple layers, perfect continuity, and regular morphology.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Canullo L, Donato A, Savadori P, Radovanovic S, Iacono R, Rakic M. Effect of argon plasma abutment activation on soft tissue healing: RCT with histological assessment. Clin Implant Dent Relat Res. 2024 Feb;26(1):226-236. doi: 10.1111/cid.13286. Epub 2023 Oct 18. PMID 37853303